CLINICAL TRIAL: NCT07160374
Title: Transarterial Drug-Eluting Chemoembolization for HCC Patients in Korea Using Transradial Approach
Brief Title: ThinkRadial: A Prospective Study of Transradial deTACE in HCC Patients
Acronym: ThinkRADIAL
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jihoon Kim, Professor, Department of Radiology, Asan Medical Center
Other Study IDs: 2017-1433
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Transarterial Chemoembolization; Drug-Eluting Beads; Transradial Access; HepaSphere; mRECIST
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transradial drug-eluting beadsTransarterial Chemoembolization (DEB-TACE) group: Patients with hepatocellular carcinoma (HCC) who undergo transarterial chemoembolization (TACE) using a transradial arterial approach with HepaSphere microspheres. Participants will be observed prospectively to evaluate the technical success, safety, and tumor response following treatment.
  Interventions: Procedure: Transradial drug-eluting beadsTransarterial Chemoembolization (DEB-TACE)

INTERVENTIONS:
Procedure: Transradial drug-eluting beadsTransarterial Chemoembolization (DEB-TACE) — Transarterial chemoembolization performed through the radial artery using HepaSphere drug-eluting microspheres in patients with hepatocellular carcinoma.

SUMMARY:
This study is a prospective, observational clinical trial designed to evaluate the feasibility, safety, and effectiveness of performing transarterial chemoembolization (TACE) for hepatocellular carcinoma (HCC) using a transradial arterial approach. Traditionally, TACE procedures are performed through the femoral artery in the groin, but using the radial artery in the wrist may reduce complications, improve patient comfort, and allow for faster recovery.

In this study, eligible patients with unresectable HCC who meet the inclusion criteria-such as preserved liver function (Child-Pugh A), good performance status, and tumors of a certain size and number-will undergo TACE using HepaSphere drug-eluting embolic materials via radial access. No randomization or drug intervention will be assigned by protocol, as the treatment will follow standard clinical practice.

The study will follow participants for 12 months to assess technical success, tumor response using imaging criteria (mRECIST), safety outcomes including adverse events, and overall survival. The study is being conducted at Asan Medical Center in Seoul, Korea, and has received Institutional Review Board approval.

DETAILED DESCRIPTION:
This is a prospective observational study to evaluate the feasibility, safety, and tumor response of transarterial chemoembolization (TACE) using a transradial approach in patients with hepatocellular carcinoma (HCC). Eligible patients will undergo drug-eluting beads TACE via radial access and be followed for up to 12 months. The primary outcome is the technical success rate of the procedure. Secondary outcomes include survival rate, tumor response by mRECIST, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

* Age between 19 and 80 years
* Diagnosed with hepatocellular carcinoma (HCC)
* Child-Pugh class A
* ECOG performance status 0 or 1
* Tumor size between 3 and 10 cm, with 1 to 7 nodules
* Ability to provide written informed consent

Exclusion Criteria:

* Child-Pugh class B or C
* Presence of other malignancies
* CKD stage 4 or 5 (eGFR < 30 mL/min/1.73m²)
* Known allergy or contraindication to contrast media
* Pregnancy or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma treated at Asan Medical Center, Seoul, Korea.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Technical Success Rate | Immediately after the procedure
  Defined as successful completion of the planned transarterial chemoembolization (TACE) procedure using transradial access without conversion to transfemoral access.

SECONDARY OUTCOMES:
Tumor Response Rate Based on mRECIST | 1-3 months post-treatment
  Assessed using modified RECIST (mRECIST) criteria by imaging studies. Includes complete response, partial response, stable disease, or progressive disease.
Incidence of Adverse Events | Within 30 days of procedure
  Number and type of adverse events observed following the TACE procedure. Severity will be graded using CTCAE criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hoon Shin, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The shared IPD will include anonymized clinical and laboratory results collected during the trial

REFERENCES:
- [Background] Fischman AM, Swinburne NC, Patel RS. A Technical Guide Describing the Use of Transradial Access Technique for Endovascular Interventions. Tech Vasc Interv Radiol. 2015 Jun;18(2):58-65. doi: 10.1053/j.tvir.2015.04.002. Epub 2015 Apr 11. PMID 26070616